CLINICAL TRIAL: NCT01371565
Title: Compassionate Use Protocol for the Administration of CORLUX® (Mifepristone) in the Treatment of the Signs and Symptoms of Endogenous Cushing's Syndrome
Brief Title: Compassionate Use of CORLUX® (Mifepristone) in the Treatment of Signs and Symptoms of Endogenous Cushing's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1073-405
Record Dates: First submitted 2011-06-07; First posted 2011-06-13 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-02

CONDITIONS: Cushing's Disease; Cushing's Syndrome
Keywords: Cushing's Disease; Cushing's Syndrome; Cushings; Pituitary; Ectopic ACTH secretion
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Cushing Syndrome; Pituitary Diseases; ACTH Syndrome, Ectopic | interventions — Mifepristone; Corlux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mifepristone (Experimental)
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — mifepristone at doses from 300mg/day up to 1200mg/day
  Other Names: CORLUX®

SUMMARY:
This is a compassionate use study. In addition to providing compassionate use access to mifepristone, objectives of the study will be to evaluate the safety and utility of mifepristone in the treatment of the signs and symptoms of endogenous Cushing's syndrome when given on a compassionate use basis. The study will only enroll subjects whose physicians have determined that medical treatment is needed to control the symptoms or signs of hypercortisolemia.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed diagnosis of endogenous hypercortisolemia caused by ACTH dependent or ACTH independent etiologies including:

   * Cushing's Disease that (more than one may apply)

     * has recurred after primary pituitary surgery
     * has persisted despite pituitary surgery (failed pituitary surgery)
     * has been treated with radiation therapy to the pituitary
     * is not treatable with surgery
     * exists in subjects who are not candidates for or who refuse surgery
   * Ectopic ACTH
   * Ectopic CRF secretion
   * Adrenal adenoma
   * Adrenal carcinoma
   * Adrenal autonomy
2. Have documented biochemical evidence of endogenous hypercortisolemia which includes elevated urinary free cortisol.
3. Require medical treatment of hypercortisolemia.

Exclusion Criteria:

Individuals not eligible to be enrolled into the study are those who:

* Have de novo Cushing's disease and are surgical candidates for pituitary surgery.
* Have an acute or unstable medical problem, which could be aggravated by mifepristone treatment.
* Taking medications within 14 days of the baseline visit (Day 1) that a) have a large first pass metabolism largely mediated by CYP3A4 and a narrow therapeutic margin and/or b) are strong CYP3A4 inhibitors.
* Female patients of reproductive potential, who are pregnant or who are unable or unwilling to use medically acceptable, non-hormonal methods of contraception during the study.
* Have received investigational treatment (drug, biological agent or device) within 30 days of Screening
* Have a history of an allergic reaction or intolerance to CORLUX (mifepristone)
* Have a non-endogenous source of hypercortisolemia such as factious hypercortisolemia (exogenous source of glucocorticoid, iatrogenic Cushing's syndrome), factious or therapeutic use of ACTH
* Have Pseudo-Cushing's syndrome.
* Postmenopausal women with an intact uterus who have experienced unexplained vaginal bleeding within 12 months of Screening are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleman Gross, M.D., Study Director — Corcept Therapeutics
Locations (5):
- United States (5):
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Division of Endocrinology Diabetes and Metabolism, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were men or non-pregnant women 18 yrs or older requiring medical treatment for symptoms of endogenous Cushing's syndrome due to ectopic ACTH, adrenal tumors/adrenal hyperplasia, or Cushing's disease if not candidates for pituitary surgery. Pts w/de novo Cushing's disease who were candidates for surgery were not enrolled.
Pre-assignment Details: All patients received active drug (no placebo).
Groups:
- Mifepristone: At doses from 300mg/day up to 1200mg/day
Period: Overall Study
Arm/Group | Mifepristone
Started | 4
Completed | 1
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Resection of neuroendocrine tumor | 1

BASELINE CHARACTERISTICS:
Population: Subjects who received one dose of study drug were included in the safety analysis.
Arm/Group | Mifepristone
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety was assessed at all visits and adverse events were recorded.
Time Frame: 6 months
Population: Due to the small number of patients enrolled (N=4), no formal assessments were planned. All patients who received study drug were included in the safety review.
Measure: Number; unit: participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 4
participants | 4

ADVERSE EVENTS:
Time Frame: From date of consent to final visit.
Description: All patients who received at least one dose of study drug are included.
Arm/Group | Mifepristone
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=4)
Adrenal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=4)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Blood potassium decreased (Investigations) | 2 (2)
Blood potassium increased (Investigations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Food craving (Metabolism and nutrition disorders) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Restless (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Jugular vein thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days